CLINICAL TRIAL: NCT01562366
Title: A Randomised, Controlled, Double-blind Clinical Investigation on the Efficacy and Safety of Radiofrequency Micro Debridement, Topaz, in Recalcitrant Greater Trochanteric Pain Syndrome (GTPS) vs. Standard of Care
Brief Title: Research Study to Compare the Addition of Topaz Micro Debridement to the Standard of Care Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SM-2012-01
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Greater Trochanteric Pain Syndrome; Hip Pain Chronic
Keywords: Iliotibial Band Release; Trochanteric Bursectomy; Micro debridement
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Device: Topaz
- Group 2 (Active Comparator)
  Interventions: Procedure: Iliotibial band release and trochanteric bursectomy

INTERVENTIONS:
Device: Topaz — Radiofrequency micro debridement with Topaz will be used to treat the gluteal tendons following standard of care procedure
  Other Names: Topaz AC-4045-01
  Arms: Group 1
Procedure: Iliotibial band release and trochanteric bursectomy — Standard of Care: An iliotibial band release and trochanteric bursectomy will be performed.
  Other Names: Standard of Care
  Arms: Group 2

SUMMARY:
Compare the surgical use of Topaz with the Standard Of Care in the treatment of Greater Trochanteric Pain Syndrome (a type of hip pain). The hypothesis is that there is a difference between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged between 40-70 years old, females and males are eligible
2. A history of > 6 months of conservative care treatment for lateral hip pain, including but not limited to local anaesthetic and steroid injections into the trochanteric bursa
3. Pre-operative MRI and ultrasound with evidence of GTPS within the previous 24 weeks
4. Willing to comply with the protocol and follow-up visits
5. Signed the Independent Ethics Committee (IEC) approved Informed Consent Form

Exclusion Criteria:

1. Previous surgery to the hip such as hip replacement, fracture neck of femur fixation, or repair of gluteal tendons
2. Subjects with sero-positive or sero-negative arthropathy
3. Long term steroid use > 6 weeks
4. Allergy to drugs to be used in the procedure
5. Medical co-morbidities that preclude surgical intervention
6. Inability to understand or respond to the study questionnaires
7. Females who are pregnant, or pregnancy is suspected or planned within the clinical investigation timeframe
8. Subjects who are simultaneously participating in another device or pharmaceutical investigation

Intra-operative Exclusion:

1. Abductor tears
2. Severe tendinopathy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Modified Harris Hip Score | 6 months
  This is a patient questionnaire used to evaluate hip function following surgery.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index | 1 year
  This is a patient questionnaire used to evaluate rheumatic symptoms, stiffness, pain and how it affects the ability to function.
Visual Analogue Scale | 1 year
  This is a patient questionnaire designed to evaluate pain.
SF-12 Health Survey | 1 year
  This is a patient questionnaire measuring health-related quality of life.
Duration of surgery between two treatment groups | 1 day
  The total length (time) of surgery will be compared between the two groups.
Ultrasound findings | 1 year
Adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John O'Donnell, M.B., B.S., Principal Investigator
Locations (1):
- Epworth Private Hospital, Richmond, Victoria, Australia

REFERENCES:
- [Derived] Blakey CM, O'Donnell J, Klaber I, Singh P, Arora M, Takla A, Fitzpatrick J. Radiofrequency Microdebridement as an Adjunct to Arthroscopic Surgical Treatment for Recalcitrant Gluteal Tendinopathy: A Double-Blind, Randomized Controlled Trial. Orthop J Sports Med. 2020 Jan 24;8(1):2325967119895602. doi: 10.1177/2325967119895602. eCollection 2020 Jan. PMID 32047828